CLINICAL TRIAL: NCT03775161
Title: A First in Human Multi-center, Open Label, Prospective Study to Evaluate the Safety, Usability and Performance of the V-LAP™ System
Brief Title: V-LAP™ Left Atrium Monitoring systEm for Patients With Chronic sysTOlic & Diastolic Congestive heaRt Failure
Acronym: VECTOR-HF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vectorious Medical Technologies Ltd. (Industry)
Collaborators: Horizon 2020 - European Commission (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CLC-0001
Record Dates: First submitted 2018-12-10; First posted 2018-12-13 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- V-LAP™ System (Experimental): Percutaneous implantation of the V-LAP™ implant by right heart catheterization (RHC) approach and daily LAP measurements at home
  Interventions: Device: V-LAP™ System

INTERVENTIONS:
Device: V-LAP™ System — Delivery of the V-LAP™ implant via a catheter-based approach in a trans-septal puncture procedure, deploying it in the inter-atrial septum.
  Other Names: Echocardiography

SUMMARY:
The purpose of the trial is to evaluate the safety, usability and performance of the V-LAP™ System in adult subjects with New York Heart Association (NYHA) Class III Heart Failure.

DETAILED DESCRIPTION:
The trial is designed to demonstrate that the V-LAP™ implant can be positioned in the interatrial septum, and that Sensor pressure measurements correlate to standardized methods of intra-cardiac pressure measurements post-sensor implant and at the 3 month follow up visit. Safety will be monitored by the occurrence of adverse events throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Ischemic or non-ischemic cardiomyopathy and documented heart failure for at least 6 months.
2. ACC/AHA Stage C, NYHA Class III or ambulatory Class IV HF documented at Baseline Visit.
3. Receiving maximally tolerated medical therapy for heart failure as indicated per ACC/AHA or ESC Heart Failure Guidelines (guideline-directed medical therapy or GDMT), such as diuretic, angiotensin-converting enzyme (ACE) inhibitor or angiotensin receptor blocker (ARB), beta-blocker (BB), and mineralocorticoid receptor blocker (MRB) for at least 3 months prior to the Baseline visit.
4. Receiving rhythm management device therapy as recommended by the ACC/AHA or ESC Guidelines. Specifically: cardiac resynchronization therapy (CRT) should be implanted for at least 90 days prior to enrollment; an implanted cardioverter-defibrillator (ICD) or a pacemaker should be implanted at least 30 days prior to enrollment. If subject is clinically contraindicated for these therapies this criterion may be waived.
5. Have a minimum of one (1) prior hospital admission within the last 12-months for acute worsening of HF associated with signs/symptoms of congestion of at least one (1) calendar date change duration requiring treatment with an intravenous diuretic. If CRT device previously implanted, the heart failure hospitalization must be ≥ 30 days after CRT implantation. Alternatively, if patients have not had a HF hospitalization within the prior 12-months, they must have a corrected* elevated Brain Natriuretic Peptide (BNP) level of at least 300pg/ml or an N-terminal pro-BNP (NT-proBNP) level of at least 1,500pg/ml, according to local measurement, within 30-days of the Baseline Visit. *Thresholds for NT-proBNP will be corrected for body mass index (BMI) using a 4% reduction per BMI unit over 20 kg/m2, If patient is on ARNI, NT-proBNP should be used exclusively.
6. Provide informed consent for study participation and be willing and able to comply with the required tests, treatment instructions and follow-up visits.

   -

Exclusion Criteria:

1. Age <18 or >85 years old.
2. Patients who are NYHA class IV not ambulatory and ACC stage D.
3. Patients with evidence/history of an intra-cardiac thrombus or history of stroke, transient ischemic attack, systemic or pulmonary thromboembolism, deep vein thrombosis (DVT), within the last 6 months.
4. Patients with a resting systolic blood pressure <90 or >180 mmHg and/ or Severe pulmonary hypertension with a pulmonary artery systolic pressure of ≥70 mm/Hg on screening baseline echocardiogram.
5. Left ventricular end-diastolic diameter (LVEDD) > 8cm.
6. Have an atrial septal defect or patent foramen ovale with more than trace shunting on color Doppler or intravenous bubble study or surgical or interventional correction of congenital heart disease involving atrial septum including placement of a PFO or ASD closure device and have a hypermobile septum or a septal aneurysm
7. Patients with untreated severe valve lesions, which are indicated for surgical or percutaneous intervention, severe regurgitant (grade 4+) valve lesions, active valvular vegetations, atrial myxoma, hypertrophic cardiomyopathy with significant resting or provoked subaortic gradient, acute myocarditis, tamponade, or large pericardial effusion, constrictive pericarditis, infiltrative cardiomyopathy (including cardiac sarcoidosis, amyloidosis, and hemochromatosis), or congenital heart disease, as cause of HF.
8. Uncontrolled tachyarrhythmia or bradycardia (heart rate <45).
9. Intractable HF with resting symptoms despite maximal medical therapy (ACC/AHA HF Stage D), including patients receiving continuous or intermittent outpatient IV vasoactive medications (e.g., IV inotropes, IV vasodilators), patients treated with a ventricular assist device (VAD).
10. Intolerant to diuretics, ACEI and ARB and beta-blocker medical therapy for patients classified as HFrEF (EF ≤40%).
11. The presence of an acute coronary syndrome (ACS), percutaneous coronary intervention (PCI), rhythm management system revision, lead extraction, or cardiac or other major surgery within the preceding 90 days.
12. Patients not eligible for emergency open-heart, thoracic or vascular surgery.
13. Women of childbearing age
14. Patients with a life expectancy that is shorter than 12 months, or those who have received a cardiac transplant or are listed for cardiac transplantation and likely to be transplanted within 12 months.
15. Have coagulopathy or uninterruptible anticoagulation therapy or contraindication for all of the forms of antiplatelet/anticoagulant treatments anticipated in the protocol
16. Have an estimated glomerular filtration rate <25 ml/min/1.73 m2 by the MDRD method or on dialysis.
17. Hepatic impairment with at least one liver Function Test (transaminases, total bilirubin, or alkaline phosphatase) ≥ 3 times upper limit of normal.
18. Gastrointestinal bleeding in the last 6 months
19. Have severe chronic pulmonary disease requiring continuous home oxygen, chronic oral steroid therapy, hospitalization for exacerbation during prior 6 months, or has severe obstructive physiology on PFTs (FEV1/FVC <0.70 and FEV1 < 50% normal).
20. Patients who have an active infection requiring systemic antibiotics or an elevated white blood count (above the local laboratory reference ranges)
21. Have a history of active drug addiction, active alcohol abuse, or psychiatric hospital admission for psychosis within the prior 2 years.
22. Are currently participating in a clinical investigation that includes an active treatment arm.
23. Subject otherwise not appropriate for study as determined by the investigator. The reasons must be documented.
24. Patients contraindicated for trans-septal puncture, TEE or ICE.

    Intra Procedural Exclusion Criteria:

    (Intra Procedural Exclusion Criteria will be determined immediately after intracardiac echocardiography or transesophageal echocardiography determination of left atrial anatomy and just before trans-septal puncture)
25. Anatomical anomaly on TEE or ICE that precludes implantation of the V-LAPIM across the interatrial septum (Fossa Ovalis) including: Septal thickness at fossa > 5 mm, FO Dimension <16mm, ASD or PFO with more than a trace amount of shunting, Intra- cardiac thrombus felt to be acute and not present on prior exams and Abnormal septum, e.g. a hypermobile septum or a septal aneurysm.
26. Inadequate vascular access for implantation of V-LAPIM or are unable to tolerate an RHC.
27. Hemodynamic at time of Index Procedure including: Severe pulmonary hypertension defined as PASP>70 mmHg or PVR >4.0 Woods Units (mmHg L-1 min-1); Resting systolic Blood Pressure <90 or >180 mmHg, not corrected with IV fluid administration or vasodilators, respectively.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-01-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Usability of the Delivery System | Intraoperative (Implantation)
  Ability to successfully deliver (to the interatrial septum) and deploy the V-LAPIM using the V-LAPDL and acutely perform initial pressure measurement.
Safety Endpoint: Study (Device and/ or system) related Major Adverse Cardiac and Neurological Events (MACNE) | Up to three months post-procedure
  (as defined in the protocol), as by the independent Clinical Events Committee

SECONDARY OUTCOMES:
Performance communication | Up to three months post-procedure
  Freedom from failure of the V-LAP system to obtain the left atrial pressure (LAP) measurement from the sensory implant and transmit the LAP data to the V-LAP Data Display
Performance accuracy | At index (baseline) and at three months
  LAP accuracy validation, concordance of the V-LAP implant measurement with pulmonary capillary wedge pressure (PCWP) measurement
Usability Assessment | Up to 24 months post procedure
  Usability Assessment of the V-LAP system will be measured by questionnaires that will be completed by the investigator, patient and medical team.

OTHER OUTCOMES:
NYHA functional class | Up to 24 months post procedure
  Change in NYHA functional class ranking during the study compare to baseline
KCCQ score | Up to 24 months post procedure
  Change in KCCQ score at 6, 12 and 24 months vs. baseline.
Heart failure hospitalization rate | Up to 60 months post procedure
  Heart failure hospitalization rate at 6, 12, 24, 36, 48, and 60 months (rate is calculated as the number of hospitalizations over individual patient follow-up duration).

CONTACTS AND LOCATIONS:
Overall Officials: Horst Sievert, Prof. Dr., Principal Investigator — Director and Founder of CardioVasculäres Centrum Frankfurt; Carlo Di Mario, Professor, Principal Investigator — University of Florence and Careggi University Hospital; Francisco Leyva, Professor, Principal Investigator — Consultant Cardiologist, Queen Elizabeth Hospital
Locations (2):
- CardioVasculäres Centrum Frankfurt, Frankfurt, Germany
- Careggi University Hospital Trust, Florence, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] D'Amario D, Meerkin D, Restivo A, Ince H, Sievert H, Wiese A, Schaefer U, Trani C, Bayes-Genis A, Leyva F, Whinnett ZI, Di Mario C, Jonas M, Manhal H, Amat-Santos IJ, Del Trigo M, Gal TB, Avraham BB, Hasin T, Feickert S, D'Ancona G, Altisent OA, Koren O, Caspi O, Abraham WT, Crea F, Anker SD, Kornowski R, Perl L; VECTOR-HF Trial Investigators. Safety, usability, and performance of a wireless left atrial pressure monitoring system in patients with heart failure: the VECTOR-HF trial. Eur J Heart Fail. 2023 Jun;25(6):902-911. doi: 10.1002/ejhf.2869. Epub 2023 May 10. PMID 37092287
- [Derived] D Ancona G, Murero M, Feickert S, Kaplan H, Oner A, Ortak J, Ince H. Implantation of an Innovative Intracardiac Microcomputer System for Web-Based Real-Time Monitoring of Heart Failure: Usability and Patients' Attitudes. JMIR Cardio. 2021 Apr 21;5(1):e21055. doi: 10.2196/21055. PMID 33881400
- [Derived] D'Amario D, Restivo A, Canonico F, Rodolico D, Mattia G, Francesco B, Vergallo R, Trani C, Aspromonte N, Crea F. Experience of remote cardiac care during the COVID-19 pandemic: the V-LAP device in advanced heart failure. Eur J Heart Fail. 2020 Jun;22(6):1050-1052. doi: 10.1002/ejhf.1900. Epub 2020 Jun 26. No abstract available. PMID 32431021